CLINICAL TRIAL: NCT00754000
Title: The AIM Study: Assessing the Impact of Margin Reduction
Acronym: AIM
Status: Completed | Type: Observational
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CMT-03-08
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: All patients in study
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — AE monitoring and EPIC QOL survey
  Other Names: EPIC survey

SUMMARY:
This study will observe patients who receive external beam radiation for prostate cancer. These patients will be localized and tracked (targeted) with the Calypso 4D Localization System. These patients will have a uniform treatment plan with reduced PTVs (prostate treatment volume) and will be assessed at multiple time points for quality of life and side effects related to radiation therapy.

DETAILED DESCRIPTION:
EPIC surveys and adverse events recorded and categorized using the CTCAE v3.0 will be collected and summary statistics performed. The patient's individual tracking graphs will be evaluated for motion type and frequency.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are planning to receive external beam radiation of prostate
2. Patients who are to be implanted with Beacon Transponders in the prostate
3. 18 years of age or older.
4. Histologically confirmed diagnosis of prostate cancer.
5. Ability to comply with study visit schedule.
6. Signed informed consent form.

Exclusion Criteria:

1. Any patients who have received other investigational therapy within the last 60 days are excluded.
2. Individuals that have previously been implanted with permanent Beacon transponders are excluded.
3. Patients that have any prosthetic implants in the pelvic region that contain metal or conductive materials (e.g., an artificial hip).
4. Any other medical or other condition that would, at the discretion of the investigator, preclude the individual from participation in a clinical study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males diagnosed with prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2008-07; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Evaluate patient quality of life using Expanded Prostate Cancer Index Composite (EPIC) for evaluation of the QOL | 2 year follow-up

SECONDARY OUTCOMES:
Collection of patient tracking data from the Calypso 4D Localization System | 9 weeks
Record the number of interventions patients receive during radiation delivery to maintain the target within the treatment plan | 9 weeks
Evaluate the user satisfaction with the Calypso 4D Localization System | At time of use
Evaluate acute and chronic (up to 2 years) toxicities of external beam prostate radiation using Common Terminology Criteria for Adverse Events for standardization of acute and chronic toxicities from the subject | 2 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Constantine Mantz, MD, Principal Investigator — GenesisCare USA
Locations (4):
- United States (4):
  - 21st Century Oncology - Scottsdale, Scottsdale, Arizona
  - 21st Century Oncology - Santa Monica, Santa Monica, California
  - 21st Century Oncology, Cape Coral, Florida
  - 21st Century Oncology - Plantation, Plantation, Florida

REFERENCES:
- [Background] Pollack A. "The Prostate" in Radiation Oncology: Rationale, Techniques and Results edited by Cox and Ang. Mosby 2003 p 630.
- [Background] Hanks GE, Leibel SA, Krall JM, Kramer S. Patterns of care studies: dose-response observations for local control of adenocarcinoma of the prostate. Int J Radiat Oncol Biol Phys. 1985 Jan;11(1):153-7. doi: 10.1016/0360-3016(85)90374-8. PMID 3967982
- [Background] Zelefsky MJ, Fuks Z, Hunt M, Yamada Y, Marion C, Ling CC, Amols H, Venkatraman ES, Leibel SA. High-dose intensity modulated radiation therapy for prostate cancer: early toxicity and biochemical outcome in 772 patients. Int J Radiat Oncol Biol Phys. 2002 Aug 1;53(5):1111-6. doi: 10.1016/s0360-3016(02)02857-2. PMID 12128109
- [Background] Zietman AL, DeSilvio ML, Slater JD, Rossi CJ Jr, Miller DW, Adams JA, Shipley WU. Comparison of conventional-dose vs high-dose conformal radiation therapy in clinically localized adenocarcinoma of the prostate: a randomized controlled trial. JAMA. 2005 Sep 14;294(10):1233-9. doi: 10.1001/jama.294.10.1233. PMID 16160131
- [Background] Chandra A, Dong L, Huang E, Kuban DA, O'Neill L, Rosen I, Pollack A. Experience of ultrasound-based daily prostate localization. Int J Radiat Oncol Biol Phys. 2003 Jun 1;56(2):436-47. doi: 10.1016/s0360-3016(02)04612-6. PMID 12738318
- [Background] Michalski JM, Purdy JA, Winter K, Roach M 3rd, Vijayakumar S, Sandler HM, Markoe AM, Ritter MA, Russell KJ, Sailer S, Harms WB, Perez CA, Wilder RB, Hanks GE, Cox JD. Preliminary report of toxicity following 3D radiation therapy for prostate cancer on 3DOG/RTOG 9406. Int J Radiat Oncol Biol Phys. 2000 Jan 15;46(2):391-402. doi: 10.1016/s0360-3016(99)00443-5. PMID 10661346
- [Background] Rudat V, Schraube P, Oetzel D, Zierhut D, Flentje M, Wannenmacher M. Combined error of patient positioning variability and prostate motion uncertainty in 3D conformal radiotherapy of localized prostate cancer. Int J Radiat Oncol Biol Phys. 1996 Jul 15;35(5):1027-34. doi: 10.1016/0360-3016(96)00204-0. PMID 8751412
- [Background] Antolak JA, Rosen II, Childress CH, Zagars GK, Pollack A. Prostate target volume variations during a course of radiotherapy. Int J Radiat Oncol Biol Phys. 1998 Oct 1;42(3):661-72. doi: 10.1016/s0360-3016(98)00248-x. PMID 9806528
- [Background] Little DJ, Dong L, Levy LB, Chandra A, Kuban DA. Use of portal images and BAT ultrasonography to measure setup error and organ motion for prostate IMRT: implications for treatment margins. Int J Radiat Oncol Biol Phys. 2003 Aug 1;56(5):1218-24. doi: 10.1016/s0360-3016(03)00290-6. PMID 12873664
- [Background] Smitsmans MH, de Bois J, Sonke JJ, Betgen A, Zijp LJ, Jaffray DA, Lebesque JV, van Herk M. Automatic prostate localization on cone-beam CT scans for high precision image-guided radiotherapy. Int J Radiat Oncol Biol Phys. 2005 Nov 15;63(4):975-84. doi: 10.1016/j.ijrobp.2005.07.973. PMID 16253772
- [Background] Litzenberg DW, Balter JM, Hadley SW, Sandler HM, Willoughby TR, Kupelian PA, Levine L. Influence of intrafraction motion on margins for prostate radiotherapy. Int J Radiat Oncol Biol Phys. 2006 Jun 1;65(2):548-53. doi: 10.1016/j.ijrobp.2005.12.033. Epub 2006 Mar 20. PMID 16545919
- [Background] Balter JM, Wright JN, Newell LJ, Friemel B, Dimmer S, Cheng Y, Wong J, Vertatschitsch E, Mate TP. Accuracy of a wireless localization system for radiotherapy. Int J Radiat Oncol Biol Phys. 2005 Mar 1;61(3):933-7. doi: 10.1016/j.ijrobp.2004.11.009. PMID 15708277
- [Background] Litzenberg DW, Willoughby TR, Balter JM, Sandler HM, Wei J, Kupelian PA, Cunningham AA, Bock A, Aubin M, Roach M 3rd, Shinohara K, Pouliot J. Positional stability of electromagnetic transponders used for prostate localization and continuous, real-time tracking. Int J Radiat Oncol Biol Phys. 2007 Jul 15;68(4):1199-206. doi: 10.1016/j.ijrobp.2007.03.030. Epub 2007 May 21. PMID 17513060
- [Background] Trotti A, Colevas AD, Setser A, Rusch V, Jaques D, Budach V, Langer C, Murphy B, Cumberlin R, Coleman CN, Rubin P. CTCAE v3.0: development of a comprehensive grading system for the adverse effects of cancer treatment. Semin Radiat Oncol. 2003 Jul;13(3):176-81. doi: 10.1016/S1053-4296(03)00031-6. PMID 12903007
- [Background] Wei JT, Dunn RL, Litwin MS, Sandler HM, Sanda MG. Development and validation of the expanded prostate cancer index composite (EPIC) for comprehensive assessment of health-related quality of life in men with prostate cancer. Urology. 2000 Dec 20;56(6):899-905. doi: 10.1016/s0090-4295(00)00858-x. PMID 11113727
- [Background] Sanda MG, Dunn RL, Michalski J, Sandler HM, Northouse L, Hembroff L, Lin X, Greenfield TK, Litwin MS, Saigal CS, Mahadevan A, Klein E, Kibel A, Pisters LL, Kuban D, Kaplan I, Wood D, Ciezki J, Shah N, Wei JT. Quality of life and satisfaction with outcome among prostate-cancer survivors. N Engl J Med. 2008 Mar 20;358(12):1250-61. doi: 10.1056/NEJMoa074311. PMID 18354103